CLINICAL TRIAL: NCT06927895
Title: Patient-Centered Care-Improving the Patient Experience in the Management of Adverse Events (AEs) Associated With Antibody Drug Conjugates (ADCs)
Brief Title: Breast Cancer Implementation Science Study With Educational Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Daiichi Sankyo (Industry); Kaplan North America (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-00449
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult Patients with HER2+/HER2 Low Breast Cancer (Experimental): Participants will receive the following educational interventions:
  1. Shared Decision Making (SDM) training video
  2. Simulation case role play (patient-clinician interactions) training video
  3. HER2-targeted ADC adverse effects and their management training video
  Interventions: Behavioral: Educational Intervention
- Clinicians in the Oncology Breast Department (Experimental): Participants will receive the following educational interventions:
  1. Shared Decision Making (SDM) training video
  2. Simulation case role play (patient-clinician interactions) training video
  3. HER2-targeted ADC adverse effects and their management training video
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — The research-specific educational intervention is the enhancement of communications and SDM in AE management.
  To this end, interventions will include pre-recorded videos that address:
  1. SDM methodologies (~30 minutes)
  2. Simulated case role play interactions between a standardized patient actor and clinician participant (~60 minutes)
  3. In depth presentation on AEs associated with HER2-targeted ADC treatments, and the management of these AEs (~45 minutes)
  Clinician participant educational intervention videos and patient participant educational intervention videos will be slightly different, as they are each presented from their specific perspectives.

SUMMARY:
A study uniquely focused on system-based practice change, measuring the impact of educational interventions on both patients and clinicians for the recognition and management of treatment-related adverse effects for HER2+/HER2 low breast cancer patients on or about to start on HER2 targeted antibody drug conjugates (fam-trastuzumab deruxtecan-nxki or ado-trastuzumab emtansine) and shared decision-making methodologies to improve adverse event (AE) management and patient-clinician communications.

ELIGIBILITY:
Inclusion Criteria, PATIENT participant group:

* ≥ 18 years of age
* Confirmed diagnosis of HER2+ or HER2 low breast cancer who are receiving or are about to receive HER2-targeted antibody drug conjugates (ADCs)
* Patient must be able to sign informed consent and be willing to participate in and comply with protocol requirements (3 visits [can be virtual], entry of survey information, access training, subset: 2 interviews and focus group) [All Virtual]
* Patient must be able to read, speak, and understand English
* Access to or ability to 1) enter information on computer or iPad into HIPAA-compliant Intelligent Dashboard online database; and 2) access training on computer or iPad

Inclusion Criteria, CLINICIAN participant group:

* Clinician agrees to see their own patients at study visits (baseline, interim time point, and end of study) in order to reduce inter-clinician variability that can affect result findings (observe effect of clinician's education on their patients' learning.)
* Clinician is a physician, NP, physician assistant, nurse, or pharmacist who works with patients with HER2-positive or HER2-low breast cancer.
* Clinician must be willing to participate in and comply with protocol requirements and provide informed consent (per IRB requirements), including availability for interviews (3), case role plays (3), patient visits (3/patient), and training
* Clinician agrees to access virtual online training videos: SDM, simulation case role play, management of adverse events for patients receiving HER2-targeted ADCs for HER2-positive or HER2-low breast cancer

Exclusion Criteria, PATIENT participant group:

* History of noncompliance
* Inability to make required "office visits" (in-person or virtual)
* Inability to participate in training
* Non-ambulatory
* Limiting comorbidities (eg. psychiatric diagnosis; significant cognitive impairment limiting ability to fulfill protocol requirements)
* Pregnant patients
* No internet and computer access

Exclusion Criteria, CLINICIAN participant group:

• Inability to participate in required virtual visits, training, assessments, and other protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) Score | Baseline
  16-item assessment of a person's uncertainty in making a healthcare choice. Each item is rated on a 5-point Likert scale from 0 (strongly agree) to 4 (strongly disagree). The total score is the sum of responses and ranges from 0-64; lower scores indicate less uncertainty. Assessed among patients only.
Decisional Conflict Scale (DCS) Score | Month 3
  16-item assessment of a person's uncertainty in making a healthcare choice. Each item is rated on a 5-point Likert scale from 0 (strongly agree) to 4 (strongly disagree). The total score is the sum of responses and ranges from 0-64; lower scores indicate less uncertainty. Assessed among patients only.
Decisional Conflict Scale (DCS) Score | Month 6
  16-item assessment of a person's uncertainty in making a healthcare choice. Each item is rated on a 5-point Likert scale from 0 (strongly agree) to 4 (strongly disagree). The total score is the sum of responses and ranges from 0-64; lower scores indicate less uncertainty. Assessed among patients only.
Patient HER2-Targeted ADC Related Side Effect Pre-Test Score | Baseline
  6 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 4 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-4 and (b) responses to items 5-6. The total score ranges from 2-14; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.
Patient HER2-Targeted ADC Related Side Effect Post-Test Score | Month 3
  6 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 4 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-4 and (b) responses to items 5-6. The total score ranges from 2-14; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.
Patient HER2-Targeted ADC Related Side Effect Post-Test Score | Month 6
  6 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 4 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-4 and (b) responses to items 5-6. The total score ranges from 2-14; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.
Clinician HER2-Targeted ADC Related Side Effect Pre-Test Score | Baseline
  7 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 5 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-5 and (b) responses to items 6-7. The total score ranges from 2-15; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.
Clinician HER2-Targeted ADC Related Side Effect Post-Test Score | Month 3
  7 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 5 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-5 and (b) responses to items 6-7. The total score ranges from 2-15; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.
Clinician HER2-Targeted ADC Related Side Effect Post-Test Score | Month 6
  7 questions assessing ability to recognize HER2-targeted ADC-related AEs and how they are managed. 5 items are multiple choice questions with (1) correct answer. The final 2 items are rated on a Likert scale from 5 (Always) to 1 (Never). The score is calculated as the sum of (a) total correct answers to items 1-5 and (b) responses to items 6-7. The total score ranges from 2-15; higher scores indicate greater ability to recognize HER2-targeted ADC-related AEs and how they are managed.

SECONDARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease Score | Baseline
  6-item assessment of a person's confidence in performing different tasks with a chronic disease. Each item is rated on a Likert scale from 1 (not at all confident) to 10 (completely confident). The score is calculated as the average of responses; the total score ranges from 1-10; higher scores indicate greater self-efficacy in managing chronic disease. Assessed among patients only.
Self-Efficacy for Managing Chronic Disease Score | Month 3
  6-item assessment of a person's confidence in performing different tasks with a chronic disease. Each item is rated on a Likert scale from 1 (not at all confident) to 10 (completely confident). The score is calculated as the average of responses; the total score ranges from 1-10; higher scores indicate greater self-efficacy in managing chronic disease. Assessed among patients only.
Self-Efficacy for Managing Chronic Disease Score | Month 6
  6-item assessment of a person's confidence in performing different tasks with a chronic disease. Each item is rated on a Likert scale from 1 (not at all confident) to 10 (completely confident). The score is calculated as the average of responses; the total score ranges from 1-10; higher scores indicate greater self-efficacy in managing chronic disease. Assessed among patients only.
Patient Satisfaction Assessment Score | Month 3
  4-item assessment of patient satisfaction with the program. Each item is rated on a scale from 0-100; the total score is the average of responses and ranges from 0-100; higher scores indicate greater patient satisfaction.
Patient Satisfaction Assessment Score | Month 6
  4-item assessment of patient satisfaction with the program. Each item is rated on a scale from 0-100; the total score is the average of responses and ranges from 0-100; higher scores indicate greater patient satisfaction.
Clinician Satisfaction Assessment Score | Month 3
  1-item assessment of clinician satisfaction with the program. The item is rated on a scale from 0-100; the total score is the item response and ranges from 0-100; higher scores indicate greater clinician satisfaction.
Clinician Satisfaction Assessment Score | Month 6
  1-item assessment of clinician satisfaction with the program. The item is rated on a scale from 0-100; the total score is the item response and ranges from 0-100; higher scores indicate greater clinician satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing Individual Participant Data, deidentified or otherwise, with any other researchers. The study design includes only deidentified, aggregate reporting.